CLINICAL TRIAL: NCT04266782
Title: ParKinWalk: Physical Activity and Long Group-walking for Motor Impairment and Quality of Life in Parkinson's Disease
Brief Title: ParKinWalk: Physical Activity and Long Group-walking for Parkinson's Disease
Acronym: ParKInWalk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Andrea Pilotto, Principal Investigator, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19/03
Record Dates: First submitted 2020-02-05; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease; Healthy Aging
MeSH Terms: conditions — Parkinson Disease | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: A group of Parkinson´s disease Patientserform physical acitivy training for three months followed by long-walking while a parallel group of PD patients will not be included in the training.
  A group of age-matched controls will be included in the training protocol as well. matched with
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinician and outcome assessors at the beginning and after the training/no intervention will not have access to the assigned arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical exercise program and Long-walking (Experimental): A physical training will be started three months before the long-walking. The subjects will have to walk for at least 3 hours per week up to 6 hours per week during the training. THe long-distance capacity will be verified in 3 different one-day walking of 10, 15 and 18 Km before the long-walking performance.
  The long-walking will be organized with the support of a physician, study nurse, physiotherapy with car support in case of need. The subject are request to complete the walk of 104 Km of Portuguese route of Santiago de Compostela walk.
  Interventions: Other: Exercise program followed by long walk in group
- Usual care (No Intervention): The subjects will be followed according to current standard.
- Control group-intervention (Active Comparator): A physical training will be started three months before the long-walking. The subjects will have to walk for at least 3 hours per week up to 6 hours per week during the training. THe long-distance capacity will be verified in 3 different one-day walking of 10, 15 and 18 Km before the long-walking performance.
  The long-walking will be organized with the support of a physician, study nurse, physiotherapy with car support in case of need. The subject are request to complete the walk of 104 Km of Portuguese route of Santiago de Compostela walk.
  Interventions: Other: Exercise program followed by long walk in group (controls)

INTERVENTIONS:
Other: Exercise program followed by long walk in group — The subjects will be included in a training exercise program for three months followed by a long-walk in group
  Arms: Physical exercise program and Long-walking
Other: Exercise program followed by long walk in group (controls) — The controls matched for age will perform the same exercise program and long walk as the PD subjects
  Arms: Control group-intervention

SUMMARY:
The study will evaluate the impact of exercise training program followed by long-walking onon supervised and unsupervised gait assessment in Parkinson´s disease and control subjects.

DETAILED DESCRIPTION:
Background: Several studies suggest an impact of physical exercise on walking parameters in Parkinson´s disease (PD) patients.

Objective: the present study will evaluate the impact of three months physical exercise training program followed by a group-long walking on motor impairment in PD.

Methods:

PD patients will be randomized in two arms: one group will be assessed to a training exercise program of three months followed by long-walking in group under the support of physician/physiotherapist and caregivers. A complete motor, cognitive and general assessment will be performed at baseline. The patients will be evaluated under supervised an unsupervised conditions at baseline, before the long-walking, during the walking and after 2 months after the walk.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson´s disease diagnosis
* stable dopaminergic treatment ( stable dose in the last three months before baseline evaluation)

Exclusion Criteria:

* gait impairment due to other medical conditions
* dementia
* impulsive compulsive disorder
* severe depression

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Supervised gait performance normal gait | Changes between baseline, immediately before the long-walking, during the day 1 and day 5 of walk and two months after walk In the non-active group- supervised and unsupervised assessment will be evaluated after 6 months of usual care.
  Step variability using wearing sensors technology in one-minute supervised walking (rehagait, Hasomed as wearing sensors)
unsupervised gait performance normal gait | Changes between baseline, immediately before the long-walking, during the day 1 and day 5 of walk and two months after walk. In the non-active group- supervised and unsupervised assessment will be evaluated after 6 months of usual care.
  Step variability using wearing sensors technology in one-day unsupervised walking (GaitUp Physilog sensors)
Supervised gait performance dual task gait | Changes between baseline, immediately before the long-walking, during the day 1 and day 5 of walk and two months after walk. In the non-active group- supervised and unsupervised assessment will be evaluated after 6 months of usual care.
  Step variability using wearing sensors technology in one-minute supervised dual task walking (Rehagait Hasomed as wearing sensors)

SECONDARY OUTCOMES:
Parkinson´s disease Quality of life questionnaire (PDQ-39) (0-117 points) Lower scores mean worse outcomes | Changes between baseline, immediately before the long-walking, during the day 1 and day 5 of walk and two months after walk. In the non-active group- the assessment will be evaluated at baseline and after 6 months of usual care.
  PDQ-39 will be assessed in patients
Unified parkinson´s disease Rating Scale part 3 (0-132 points) Higher scores mean worse outcomes | Changes between baseline, immediately before the long-walking, during the day 1 and day 5 of walk and two months after walk. In the non-active group- the assessment will be evaluated at baseline and after 6 months of usual care.
  Total Movement Disorder Society-Unified Parkinson's disease Rating Scale part 3 motor score

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Padovani, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Department of Neurology ASST Spedali Civili Brescia, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Wearing sensor will be available after completion of the trial
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the completion fo the trial this will be presented in a publication
Access Criteria: upon reasonable request